CLINICAL TRIAL: NCT01214382
Title: A Prospective, Longitudinal Comparison of the Pharmacokinetic Properties of Sertraline Before and After Roux-en-Y Gastric Bypass
Brief Title: Pharmacokinetic Properties of Sertraline Before and After Gastric Bypass Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: North Dakota State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Kristine Steffen, Associate Professor, North Dakota State University, Neuropsychiatric Research Institute, Fargo, North Dakota
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 1K23DK085066-01 (NIH)
Record Dates: First submitted 2010-09-30; First posted 2010-10-05 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Roux en Y Gastric Bypass Surgery
Keywords: Gastric Bypass; Bariatric Surgery; Sertraline; Zoloft; Pharmacokinetic
MeSH Terms: interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sertraline (Experimental)
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Sertraline — Single dose sertraline 100 mg, tablet and solution
  Other Names: Zoloft

SUMMARY:
This study is being conducted to evaluate how the body absorbs and processes the medication sertraline (Zoloft®) before compared to how it is absorbed at two time points after gastric bypass surgery. Participants will be asked to take part in this study at three time points: 1) before their bariatric surgery, 2) at three months following the surgery, and 3) twelve months following surgery. This study will enroll approximately 30 participants.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female between 18 and 60 years of age at the time of Informed Consent
* 2. Scheduled to undergo Roux en Y Gastric Bypass Surgery (RYGBP) or in evaluation for surgery prior to scheduling at the investigators' discretion.
* 3. Ability to swallow whole medication tablets and eat solid foods

Exclusion Criteria:

* 1. Those taking any medication at the time of the study which has a known, clinically significant, drug-interaction with sertraline, which may affect participant safety or threaten the validity of the data.
* 2. Hypersensitivity to sertraline or any excipient contained in either the tablet or solution
* 3. Inability to tolerate blood draws
* 4. History of or current bipolar disorder, psychotic disorder, or current major depressive disorder or suicidality, or other psychiatric condition that the investigator feels may put the subject at additional risk by participating in the study
* 5. Alcohol or other substance abuse in the past four weeks or dependence in the past year
* 6. Currently pregnant or lactating or any participant who wants to become pregnant during the study
* 7. Female participant unwilling to use an accepted method of birth control during the study assessment periods.
* 8. Disulfiram or metronidazole at baseline (due to small percentage of alcohol in sertraline solution) or other medication with a similar interaction with a very small amount of alcohol
* 9. Inability or unwillingness to avoid alcohol or grapefruit juice for the required study duration
* 10. Baseline medications which significantly alter gastrointestinal transit time (e.g. oral anticholinergic medications, metoclopramide, erythromycin) and are taken on a routinely scheduled basis. In addition, any such medication cannot be taken in close proximity (minimum of five half-lives of the drug) to the study sertraline administration.
* 11. Medical condition which may increase participant risk with sertraline
* 12. Hepatic insufficiency (Hepatic insufficiency will be defined as any liver enzyme test on a standard hepatic panel of greater than or equal to twice the upper limit of normal, or any other hepatic abnormality identified on physical exam, self-report, or laboratory testing that puts the participant at risk in the opinion of the study physician or physician assistant.)
* 13. History of daily tobacco product use in the past six months
* 14. Participants who have undergone any type of prior surgical procedure for weight loss
* 15. Significant Latex allergy (liquid form has a latex dropper)
* 16. Participant employed by, or who has immediate family employed by NRI
* 17. History of Hepatitis or HIV Infection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2010-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Sertraline Plasma Concentrations/Area-Under-the-Curve (AUC) | 72 hour intervals
  The primary aim of this research is to provide a prospective, longitudinal comparison of pharmacokinetic measures associated with a single-dose of sertraline in RYGBP patients. Comparisons will be based upon sertraline plasma concentrations obtained prior to surgery and repeated at three and 12 months following surgery. A 24+ month post-surgery follow-up to evaluate sertraline tablet AUC will be offered to a subset of study volunteers.

SECONDARY OUTCOMES:
Bioavailability comparison between sertraline tablet and sertraline liquid | 72 hours
  To characterize the relative bioavailability of the tablet formulation of sertraline 100mg as compared to a reference dose of the liquid preparation of sertraline 100mg before and at three and 12 months following RYGBP.
Body Composition and Weight | 72 hours
  Chanes in body compsition and weight will be correlated with changes observed in sertraline pharmacokinetic parameters and will be considered exploratory.
Hepatic Function | 72 hours
  To assess the area under the curve (AUC) ratio of N-desmethylsertraline to sertraline as a measure of hepatic function over time.
Plasma Protein Concentrations | 72 hours
  To assess changes over time in common drug binding plasma proteins in relationship to observed sertraline plasma levels.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine J Steffen, Pharm.D., Ph.D., Principal Investigator — Neuropsychiatric Research Institute
Locations (1):
- Neuropsychiatric Research Institute, Fargo, North Dakota, United States

REFERENCES:
- See also: Neuropsychiatric Research Institute Website — http://www.nrifargo.com